CLINICAL TRIAL: NCT04193358
Title: Impact of A Nutritional Supplements' Combination (FERTILIS) On Male Infertility: A Monocentric Double Blind Randomized Placebo Controlled Trial
Brief Title: Impact of A Nutritional Supplements' Combination (FERTILIS) on Male Infertility
Acronym: FERTILIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Les Laboratoires des Médicaments Stériles (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FERTILIS-349
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-03

CONDITIONS: Infertility, Male; Subfertility, Male
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Intervention Model Description: Comparative, interventional, prospective, monocentric, double blind, randomized, placebo controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FERTILIS HOMME® group (group A) (Experimental): Group A will receive 2 FERTILIS HOMME capsules twice daily to be taken with meals for 3 months.
  Interventions: Dietary Supplement: FERTILIS HOMME®
- Placebo group (group B) (Placebo Comparator): Group B will receive 2 placebo capsules twice daily to be taken with meals for 3 months
  Interventions: Other: PLACEBO

INTERVENTIONS:
Dietary Supplement: FERTILIS HOMME® — L-carnitine 220 mg, Zinc 20 mg, Selenium 0.03 mg, L-arginine 125 mg, L-glutathione 40 mg, Folic acid (vitamin B-9) 0.4 mg, Coenzyme Q10 7.5 mg, and Vitamin E 60 mg
  Arms: FERTILIS HOMME® group (group A)
Other: PLACEBO — Sugar pills
  Arms: Placebo group (group B)

SUMMARY:
Infertility is a major health problem affecting up to 15% of couples of reproductive age globally. For several years, it was assumed that most reproductive problems could be attributed to the female partner, but research in recent years has demonstrated that males were solely responsible for 20-30% of infertility cases and contributed to 50% of infertility cases overall. The term ''male infertility'' does not constitute a defined clinical syndrome, but rather a collection of different conditions exhibiting a variety of etiologies.

It is far increasingly known that reactive oxygen species (ROS) are of significant pathophysiological importance in the etiology of male infertility. ROS are highly reactive oxidizing agents belonging to the class of free radicals containing one or more unpaired electrons, which are continuously being generated through metabolic and pathophysiologic processes. It has been suggested that oxidants interfere with normal sperm function via membrane lipid peroxidation and fragmentation of nucleic acids, which result in sperm dysfunction. Due to the sperm cell membrane abundance of polyunsaturated fatty acids (PUFAs) and the capacity of sperm to generate ROS, human spermatozoa are highly susceptible to oxidative stress.

Since growing evidence indicates that oxidative stress can be a primary cause of male infertility, non-enzymatic antioxidants play a significant protective role against oxidative damages and lipid peroxidation. In addition, micronutrients and antioxidants are often used with good results in men with idiopathic infertility.

Keeping in view the main protection provided by seminal plasma antioxidants against oxidative damages, a previous study showed that the dietary management with an eight nutritional supplements' combination, similar to this study's product and containing antioxidants, achieved a significant improvement in sperm quality up to a completely normal semen analysis. Also, another study confirmed the hypothesis that the combination of individual nutritional supplements as described in literature showed significantly better results than the sum of the effects of single administration.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 20 years of age
* Attending the Department of Obstetrics and Gynecology of Farhat Hached University Hospital, Sousse, Tunisia, for consultation or semen analysis as part of infertility investigations
* Diagnosis of oligozoospermia (WHO 2010 definition)
* Diagnosis of Asthenozoospermia (WHO 2010 definition)
* Diagnosis of teratozoospermia1 (WHO 2010 definition)
* Diagnosis of idiopathic infertility
* Couple is candidate for Intrauterine Insemination (IUI), In Vitro Fertilization (IVF) and/or Intracytoplasmic Sperm Injection (ICSI).

Exclusion Criteria:

* Inclusion visit (prior to treatment initiation): Patients will be selected during this initial visit if they meet all inclusion and none of the exclusion criteria.
* Randomization visit: around 1-week post inclusion visit: Patients will be given either of study interventions.
* Follow up visit 1-month post treatment initiation: Patients will be given study interventions' refill for 1 month.
* Follow up visit 2-months post treatment initiation: Patients will be given study interventions' refill for another month.
* Follow up visit 3-months post treatment initiation: Patients will undergo laboratory assessment.
* Follow up visits every 3-months post Visit: Patients' female partner will undergo laboratory and clinical assessment.
* End of trial (CLOSING) visit 24-months post treatment initiation: Patients' female partner will undergo laboratory and clinical assessment.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Sperm DNA fragmentation Index (DFI) | 3 months
  To evaluate the effect of a nutritional supplement's combination of 8 active compounds (L-carnitine 220 mg, Zinc 20 mg, Selenium 0.03 mg, L-arginine 125 mg, L-glutathione 40 mg, Folic acid (vitamin B-9) 0.4 mg, Coenzyme Q10 7.5 mg, and Vitamin E 60 mg; FERTILIS HOMME®, Les Laboratoires MédiS, Tunisia), on sperm DNA fragmentation index (DFI).

SECONDARY OUTCOMES:
Sperm quantity | 3 months
  Ejaculatory volume (ml) and sperm cell density (mill/ml
Sperm quality | Up to 3 months
  Sperm morphology and sperm total motility/progressive motility
Occurrence of spontaneous pregnancy | Through study completion, an average of 2 years
Occurrence of pregnancy consecutive to Assisted Reproductive Technology (ART) | Through study completion, an average of 2 years
Fertilization rate during in vitro fertilization (IVF) | Up to 3 months
Embryo cleavage rate and embryo quality during intracytoplasmic sperm injection (ICSI) | Up to 3 months
Achievement of clinical pregnancy | Through study completion, an average of 2 years
Achievement of live birth | Through study completion, an average of 2 years
Number of Adverse Events | Through study completion, an average of 2 years
  To assess the safety of the study product

CONTACTS AND LOCATIONS:
Overall Officials: Mounir Ajina, Dr., Principal Investigator — Farhat Hached Hospital; Latifa Lassoued, Dr., Principal Investigator — Farhat Hached Hospital
Locations (1):
- Farhat Hached Hospital, Sousse, Tunisia